CLINICAL TRIAL: NCT06873165
Title: Development of Microbial Therapeutics for Metabolic-associated Fatty Liver Disease: From Mechanistic Investigations to Clinical Trials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 202403035RSC
Record Dates: First submitted 2025-03-06; First posted 2025-03-12 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-01

CONDITIONS: Metabolic Dysfunction-Associated Steatotic Liver Disease
Keywords: Metabolic Dysfunction-Associated Steatotic Liver Disease; Akkermansia muciniphila
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Placebo (Placebo Comparator): 1 capsule per day for 12 weeks
  Interventions: Dietary Supplement: Placebo
- Active Comparator: AKK-1 (Active Comparator): 1 capsule (with 1000000000 CFU pAKK LWHK0003) per day for 12 weeks
  Interventions: Dietary Supplement: Probiotics
- Active Comparator: AKK-2 (Active Comparator): 1 capsule (with 10000000000 CFU pAKK LWHK0003) per day for 12 weeks
  Interventions: Dietary Supplement: Probiotics
- Active Comparator: AKK-3 (Active Comparator): 1 capsule (with 100000000000 CFU pAKK LWHK0003) per day for 12 weeks
  Interventions: Dietary Supplement: Probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics — 1 capsule(with three different dosage) per day for 12 weeks
  Other Names: Akkermansia muciniphila
  Arms: Active Comparator: AKK-1; Active Comparator: AKK-2; Active Comparator: AKK-3
Dietary Supplement: Placebo — 1 capsule per day for 12weeks
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to investigate the efficacy and safety of pasteurized Akkermansia muciniphila strain NTUH_Amuc03 (pAKK NTUH_Amuc03) in Metabolic Dysfunction-Associated Steatotic Liver Disease (MASLD)Patients. The main question it aims to answer is:

Does pAKK NTUH_Amuc03 trend to reduce the body weight, improve abnormal blood lipids , NASLD activity score, and HOMA-IR ?

Researchers will compare pAKK NTUH_Amuc03 to a placebo (a look-alike substance that contains no Akk) to see if pAKK NTUH_Amuc03 works to MASLD.

Participants will:

1. Take capsule with pAKK NTUH_Amuc03 or a placebo every day for 3 months
2. Visit the clinic once every 4 weeks for checkups and tests

DETAILED DESCRIPTION:
Metabolic Dysfunction-Associated Steatotic Liver Disease(MASLD)is an improved diagnostic standard derived from Non-Alcoholic Fatty Liver Disease (NAFLD), emphasizing the correlation between fatty liver and metabolic dysfunction. Compared to NAFLD, which requires the exclusion of various conditions for diagnosis, the diagnostic criteria for MASLD can enhance the homogeneity of study subjects. It also addresses various groups with coexisting liver diseases, aiding in the efficiency and applicability of new drug development. MASLD has a prevalence rate of approximately one-fourth of the global population. If left untreated and worsens, it may lead to liver fibrosis, cirrhosis, or even liver cancer. Due to the significant medical burden associated with MASLD and the lack of FDA-approved treatments, the development of therapeutic methods for MASLD is an urgent issue. Past literature indicates that diet and gut microbiota play crucial roles in the progression of MASLD. The composition of the diet affects gut microbiota and intestinal barrier function. In cases of dysbiosis, harmful substances produced by gut microbiota, including pathogen-associated molecular patterns (PAMPs) and microbiota-dependent metabolites (MDMs), enter the liver through the portal vein via the leaky gut, resulting in toxicity. The pathogenic pathways exacerbating MASLD through gut microbiota dysbiosis, collectively termed the gut-liver axis, are not fully understood. Some animal studies have found dietary supplements to regulate gut microbiota beneficial for improving MASLD. Although most lack clinical evidence, incorporating food components that regulate gut microbiota and immune function into the diet indeed holds potential for treating MASLD. Next-generation probiotics have been found in past studies to improve liver lipid metabolism and regulate gut microbiota. They may slow the progression of MASLD by modulating the gut-liver axis. Previous studies by our team applied the pasteurized Akkermansia muciniphila strain NTUH_Amuc03 (pAKK NTUH_Amuc03), in preclinical animal studies to alleviate fatty liver disease progression. In experiments with mice induced with high-fat, high-fructose, high-cholesterol diets, pAKK NTUH_Amuc03 trended to reduce the body weight, improve abnormal blood lipids in mice, NASLD activity score, and HOMA-IR. These results indicate the potential of pAKK NTUH_Amuc03 to slow the progression of MASLD. Therefore, this project aims to further evaluate the efficacy and safety of pAKK NTUH_Amuc03 in MASLD patients through clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects aged between 20 and 70 years old.
* The subject is diagnosed through FibroScan (CAP≧ 260 db/m)and meets one of below .
* the subject's BMI ≧23 kg/m² or waist ≧ 90cm (male) 80cm (Female)
* Fasting glucose≧100 mg/dL or sugar after meal ≧140 mg/dL or HbA1c≧5.7 or diagnosed type II diabetes(including under treatment or not)
* Blood pressure≧ 130/80 mmHg or under medication.
* Blood Triglycerides≧150 mg/dL or under medication.
* Blood HDL ≤ 40 mg/dL (Male) ≤ 50 mg/dL (Female) or under medication.
* If the subject is reproductive women, she should agree to take more than two ways of contraceptive methods.
* The subject is able to provide written informed consent by himself/herself and agrees to comply with all protocol requirements.
* The subject agrees to comply with the following two requirements:

comply with all follow-up visit requirements according to the trial protocol. comply with all requirement regarding fecal samples collection, storage and delivery according to the trial protocol.

Exclusion Criteria:

* The subject is pregnant or lactating.
* The subject has received probiotics or prebiotics 14 days prior to visit 1.
* The subject has received any antibiotic (excluding topical agents) or antifungals within 30 days prior to visit 1.
* The subject has received medication affecting evaluating indicators 14 days prior to visit 1, including steroids, immunosuppressant or anti-inflammation drugs hepatitis and lipid, metabolism related compounds, but excluding the following medicines: Statins, Fibrates, Silymarin, Thiazolidinediones, Metformin, Fibrate, Cholestyramine, Ezetimibe, Orlistat, SGLT2i and GLP1-RAs.

If the above-mentioned drugs are used continuously for more than six months and the dosage is not changed during the trial,this situation is accepted.

* The subject has a clinically significant, currently active or underlying diarrhea (loose stools more than three times in 24 hours) of infectious etiologies.
* The subject who has been diagnosed a severe/injury hepatic disease, disease affecting liver function, active inflammatory bowel disease.
* Acute hepatitis caused by viruses or other causes and ALT > 200 U/L.
* Coronary artery disease with arterial stent surgery in half year.
* Fasting glucose≥ 300 mg/dl or HbA1c>9%.
* Blood triglyceride≥ 500 mg/dl.
* The subject currently is participating in studies involving other investigational drugs, medical devices, functional foods, or cosmetic within 30 days prior to visit 1.
* The subject has participated in body weight control plan within 60 days prior to visit 1.
* The subject has been aboard for 10 days within 60 days prior to visit 1, or plans to go aboard during this study.
* The subject is special diet.
* The subject is considered by the investigator as not suitable for the trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Changes in gut microbiota | baseline and after 12-13th weeks
  evaluated by fecal 16S rRNA gene sequencin
Improvement of intrahepatic fibrosis | baseline 、 12th and 16th weeks
  evaluated by FibroScan

SECONDARY OUTCOMES:
Changes in FIB-4 | baseline 、 12th and 16th weeks
  Fibrosis-4 (FIB-4) Index
Changes in gut permeability | baseline to 12th week
  evaluated by lactulose/mannitol ratio

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: The globalization of nonalcoholic fatty liver disease: Prevalence and impact on world health — https://pubmed.ncbi.nlm.nih.gov/26926530/
- See also: Metabolic risk factors are associated with non-hepatitis B non-hepatitis C hepatocellular carcinoma in Taiwan, an endemic area of chronic hepatitis B — https://pubmed.ncbi.nlm.nih.gov/29881825/
- See also: Global burden of NAFLD and NASH: trends, predictions, risk factors and prevention — https://pubmed.ncbi.nlm.nih.gov/28930295/